CLINICAL TRIAL: NCT06396247
Title: Impact of Brief Daily Functional Resistance Training on Lower Extremity Physical Performance
Acronym: FASTNIA
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Christopher Sciamanna, MD, MPH, Professor of Medicine, Penn State Health Milton S Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00024492; R01AG079938 (NIH)
Record Dates: First submitted 2024-04-29; First posted 2024-05-02 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Mobility Limitation
Keywords: older adults; walking; mobility
MeSH Terms: conditions — Mobility Limitation

STUDY DESIGN:
Intervention Model Description: We hypothesize that patients assigned to FAST will improve these outcomes significantly more than those assigned to DTC and that FAST participants with higher levels of perceived exertion and adherence will improve these measures the most.
Who Masked: Participant, Investigator
Masking Description: Randomization
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Functional Activity Strength TRaining (Experimental): Participants will perform 5 minutes of functional resistance training daily, supported by 24 video coaching sessions over 12 months.
  Interventions: Behavioral: Functional Activity Strength Training
- Delayed Treatment (Active Comparator): Participants will receive the intervention after 12 months.
  Interventions: Behavioral: Functional Activity Strength Training

INTERVENTIONS:
Behavioral: Functional Activity Strength Training — FAST consists of five exercises (stepping on a step, chair stands, push-ups, rows, walking), for 30 seconds each, performed daily, with 30 seconds of rest between.

SUMMARY:
In this study, we will randomly assign 360 older adults to 12 months of 5 minutes per day of functional resistance training or to a delayed treatment control condition, and measure the impact of the training on measures of lower extremity performance and walking ability.

DETAILED DESCRIPTION:
One of the most common, and untreated, health problems among older adults is mobility disability, observed in nearly one in five (17.9%) of older adults. Mobility disability is typically the first disability to develop and increases future risk for additional disabilities and death. Though the most effective treatments for mobility disability are forms of exercise, especially resistance training (RT), they are rarely used, with fewer than 20% of older adults meeting RT guidelines and even fewer among those with mobility disability. The core problem of disseminating the benefits of RT to older adults is adherence. One potential opportunity to enhance adherence to RT, which has not been tested, is to make RT programs shorter. Studies show that most of the benefits of RT accrue with the first few sets per week, consistent with the law of diminishing utility. While traditional RT programs for older adults, like those offered by Silver Sneakers, are typically 45 minutes three times weekly, fewer than 5% of older adults with free access to these programs participate. Our qualitative work shows that older adults often feel that 45 minute sessions are too challenging (e.g., "I don't think I have the strength to do it for 45 minutes") and 75% of older adults we surveyed preferred a 5 minute RT to a 45 minute RT option, assuming they were equally effective. In 2020, we set out to design a brief, home-based RT program that would lead to both high levels of adherence and functional improvement. We called the program FAST (Functional Activity Strength Training) and, to overcome its brevity, FAST was augmented with several standard behavior change techniques (e.g., feedback, reminders, self-monitoring) and a novel form of goal- setting, rarely used in RT studies, for the number of additional repetitions participants should be able to do during the study. In FAST-1, 24 healthy older adults were prescribed 30 seconds of squats and push-ups each day and given no personal supervision. Over 6 months, they performed the exercises on 73% of days and showed large increases in squat and push-up performance (Cohen's d > 1.0). In FAST-2, we randomly assigned 97 older adults with mobility disability, and those assigned to 30 seconds each of chair stands and steps onto a stepper each day completed exercises on 81% of days (5.7 days per week) and improved their 5 time sit-to-stand test (-2.8 seconds, Cohen's d=0.53), 30 second chair stand test (+4.2 repetitions, d=1.1) and One Leg Stand test (+3.7 seconds, d=0.40), versus controls. In this multicenter study, we will randomly assign 360 older adults with an SPPB score < 8 to 6 months of daily FAST or to a delayed control group. We will test the impact of FAST on physical performance, walking ability, falls and functional limitations. We hypothesize that FAST will improve these measures more than controls, and that those with greater adherence and perceived effort will improve the most. By rigorously testing FAST, we hope to change the paradigm of RT prescription from "More is better" to "What will people do that works?" and, if FAST proves superior, a future study will test whether FAST leads more older adults to do RT and, thereby, improve the public's health.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported difficulty or inability to walk ¼ mile

Exclusion Criteria:

* Chest pain on the PAR-Q

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2025-04-09 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Short Physical Performance Battery | Baseline, 6 months, 12 months
  The SPPB assesses balance, gait speed, and lower extremity strength.

CONTACTS AND LOCATIONS:
Overall Officials: Maggie Nellissery, Ph.D., Study Chair — National Institute on Aging (NIA)
Locations (2):
- United States (2):
  - Penn State College of Medicine, Hershey, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
We estimate the upload at 10MB, as we have experience uploading our data into ICPSR
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 12 months after study has completed
Access Criteria: ICPSR Account holder
URL: https://www.icpsr.umich.edu/web/pages/